CLINICAL TRIAL: NCT02115971
Title: The Effect of a 12-week Training Jumping Exercises Program in Individuals With Chronic Ankle Instability: Randomized Controlled Trial Pilot Study
Brief Title: Jumping Exercises Approach in Individuals With Chronic Ankle Instability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment process could not provide us with enough participants
Sponsor: Swanenburg (Other)
Responsible Party: Sponsor-Investigator, Swanenburg, PhD, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Balgrist 2009-124; KEK-ZH-Nr. 2009-124 (Other: Ethics commission of the Canton Zurich, Switzerland)
Record Dates: First submitted 2014-04-03; First posted 2014-04-16 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Joint Instability; Chronic Disease; Sprains
Keywords: chronic; functional; instability; ankle
MeSH Terms: conditions — Joint Instability; Chronic Disease; Sprains and Strains; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jumping exercise (Experimental): Physical therapy with a focus on specific jumping exercise. The jumping exercise will be performed for 12 weeks (3x/week), with a break of day between workouts. The 40-minute workout is completed 2 times under supervision in the clinic's internal training group for outpatients. 1 time they train on their own at home, based on a defined training program. The training process is documented by the training protocol.
  The incipient exercise intensity is taking personal performance into account. The exercise intensity is increased by a progressive scheme.
  Interventions: Other: Jumping exercise
- Strength exercise (Active Comparator): Physical Therapy with a focus on stability and strength exercise. Strength exercise arm has also same duration of 12 weeks with comparable intensity. The program is according to a predetermined program. The 60-minute training is completed twice under supervision in the clinic's internal training group for outpatients.There is no contact with participants of other group.
  Between the two exercise sessions there is a training free day. The training process is documented by the training protocol. The incipient exercise intensity is considering personal performance. The intensity is increased after workout usual principles. The exercises are described with clear image and load parameters. The training exercises are regularly monitored.
  Interventions: Other: Strength exercise

INTERVENTIONS:
Other: Jumping exercise — Total 120min exercise
  Arms: Jumping exercise
Other: Strength exercise — Total 120 min exercise
  Arms: Strength exercise

SUMMARY:
The aim of this pilot study is to analyze the effect of a 12-week specific jump training compared with conventional therapy in patients with chronic functional instability of the ankle. It is to be evaluated to what extent the symptoms in of chronic functional instability of the ankle can be influenced in everyday life.

DETAILED DESCRIPTION:
There is a need for;

1. more homogeneous sub- groups with chronic functional instability of the ankle.
2. Studies are needed that older patients (up to 50 years) and also take into account women.
3. In addition, studies should be performed in a clinical environment and also at the same time clinically adapted test can be used as a form measurement.

( Hiller et al. , 2011).

ELIGIBILITY:
Inclusion Criteria:

* Ankle injury more than 6 months ago
* Chronic instability
* Functional instability of the ankle
* Experience with proprioceptive exercises

Exclusion Criteria:

* Foot surgery
* Fresh ankle injury
* Acute foot pain with signs of inflammation
* Mechanical / anatomical ankle instability
* Athletes with regularly jumping exercise (eg volleyball, basketball)
* Taking medications which affect balance and coordination
* Diseases that affect the balance
* Serious diseases such as tumors, infections, neuropathies, severe articular degeneration
* Non-German-speaking patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Gait variables | Change from Baseline in Gait variables at week 3, week 7, and at the end of therapy (week 12)
  Gait variables will be assessed with the OptoGait system OptoGait system is a floor-based photocell system for measuring spatiotemporal gait parameters.
  All measurements will be executed within 1hour

SECONDARY OUTCOMES:
Balance | Baseline, week 3, week 7, and at the end of therapy (week 12)
  Time to Stability (Forceplate Accusway AMTI)
  * 1 leg jump test
  * step down test
Health questionnaire | Baseline, week 3, week 7, and at the end of therapy (week 12), followup 12 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.
Foot function questionnaire | Baseline, week 3, week 7, and at the end of therapy (week 12)
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments.
Personal calendar | 12 months
  Participant could enter any new ankle sprain into this calendar. As soon as possible after new ankle sprain the participant had to fill in the date, its cause, and sprain-related injuries. The calendar pages contained questions about the circumstances surrounding the new ankle sprain, including how and where it happened, activity performed, possible injury symptoms, time to recover and whether medical assistance or physical therapy was needed. Participants are also requested to record direct medical costs (e.g. physiotherapy, visits to general practitioners and medical specialists, nursing care, and medication) and indirect cost (e.g. disability related loss) using the "personal calendar". At the end of 2 month, a calendar page was sent by each patient to the investigators

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanneburg, PhD, Principal Investigator — Balgrist Univeresty Hospital
Locations (1):
- Balgrist Univeresty Hospital, Zurich, Canton of Zurich, Switzerland